CLINICAL TRIAL: NCT05716607
Title: Randomized Cross-over Trial in Patients Treated With Both Insulin & Hydrocortisone
Brief Title: Treatment Study in Patients Treated With Both Insulin & Hydrocortisone
Acronym: INSCORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: The Swedish Society of Medicine (Other); Åke Wibergs Stiftelse (Unknown); Sahlgrenska University Hospital (Other); Pilloxa (Industry)
Responsible Party: Principal Investigator, DimitriosChantzichristos, Principal Investigator, Vastra Gotaland Region
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INS.CORT
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Adrenal Insufficiency; Polyglandular Autoimmune Syndrome
Keywords: Insulin treatment; Hydrocortisone treatment; Opposing effects on glucose metabolism; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus; Adrenal Insufficiency; Polyendocrinopathies, Autoimmune

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, open-label, two-period cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once-daily dual-release hydrocortisone (Experimental)
  Interventions: Drug: OD dual-release Hydrocortisone
- Thrice-daily conventional immediate-release hydrocortisone (Active Comparator)
  Interventions: Drug: TID Hydrocortisone

INTERVENTIONS:
Drug: OD dual-release Hydrocortisone — Treatment with once-daily dual-release hydrocortisone
  Other Names: Once-daily dual-release hydrocortisone
  Arms: Once-daily dual-release hydrocortisone
Drug: TID Hydrocortisone — Treatment with thrice-daily conventional immediate-release hydrocortisone
  Other Names: Thrice-daily conventional immediate-release hydrocortisone
  Arms: Thrice-daily conventional immediate-release hydrocortisone

SUMMARY:
The aim of INS.CORT trial is, by studying glycemic variability in a well-defined patient group with both insulin & hydrocortisone (patients with concomitant insulin-treated diabetes & Addison's disease) and collecting information about the administration -time point and doses- of insulin, hydrocortisone and food intake with the help of new technology to improve the treatment in all patients treated with both insulin & glucocorticoids.

ELIGIBILITY:
Inclusion Criteria:

Men and women at age 18 to 70 years, with BMI 18-32 kg/m2 and well-defined both insulin-treated diabetes & Addison's disease for >12 months each, on insulin treatment and stable hydrocortisone replacement with once-daily dual-release hydrocortisone (20-30 mg/day) for >3 months.

Exclusion Criteria:

* Any medication with other glucose lowering agents than insulin
* Any additional underlying or intercurrent disease that may need regular or periodic pharmacological treatment with glucocorticoids during the study period, including infectious diseases
* Any medication with agents which in the investigator's judgement might interfere with the study drugs kinetics, including therapies affecting gastrointestinal emptying or motility
* Any medication with oral estrogen supplementation and/or regular DHEA medication for the past 4 weeks
* Clinically significant renal dysfunction with a serum creatinine above 160 mmol/L
* Active malignancy
* Clinical or laboratory signs of significant cerebral, cardiovascular, respiratory, hepatobiliary/pancreatic disease which in the investigator's judgement may interfere with the study assessment
* Pregnant or lactating women
* Alcohol/drug abuse or any other condition associated with poor patient compliance, including expected non-cooperation, as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
glycemic variability | 4 weeks
  glycemic variability

SECONDARY OUTCOMES:
HbA1c | 4 weeks
  HbA1c
Time in range (glucose) | 4 weeks
  Time in range (glucose)
Time above range (glucose) | 4 weeks
  Time above range (glucose)
Time below range (glucose) | 4 weeks
  Time below range (glucose)
Cortisol exposure-time profile | 4 weeks
  Cortisol exposure-time profile
systolic blood pressure | 4 weeks
  systolic blood pressure in sitting position
diastolic blood pressure | 4 weeks
  diastolic blood pressure in sitting position
ADDIQoL | 4 weeks
  questionnaire: the Addison-specific quality-of-life (ADDIQoL)
  The AddiQoL is a 36-item questionnaire; each item contains six scoring categories. Twenty-five items are negative Health-Related Quality of Life (HRQoL) statements that need to be reversed for questionnaire scoring; thus, a higher score indicates a higher level of HRQoL.
PGWB | 4 weeks
  questionnaire: the Psychological General Well-Being (PGWB) index
  The Psychological General Well-Being Index (PGWBI) is a measure of the level of subjective psychological well-being. In detail, it assesses self-representations of intrapersonal affective or emotional states reflecting a sense of subjective well-being or distress and thus captures what we could call a subjective perception of well-being. Consisting of 22 standardized items (6 items for the short form), the tool produces a single measure of psychological well-being. The full measure also provides sub-scales to assess the following domains: anxiety, depression, positive well-being, self-control, general health, and vitality.
FIS | 4 weeks
  questionnaire: the Fatigue Impact Scale (FIS)
  The FIS was developed to assess the symptom of fatigue as part of an underlying chronic disease or condition. Consisting of 40 items, the instrument evaluates the effect of fatigue on three domains of daily life: cognitive functioning, physical functioning, and psychosocial functioning minimum and maximum values, and whether higher scores mean a better or worse outcome.
  Higher scores mean a worse outcome. Min 0 points, max 160 points.
FOSQ | 4 weeks
  questionnaire: the Functional Outcomes of Sleep Questionnaire (FOSQ)
  Disease specific quality of life questionnaire to determine functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment. Name of categories assessed: Activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome, rate the difficulty of performing a given activity on a 4-point scale (no difficulty to extreme difficulty).
  Higher scores mean a better outcome. Min 0 points, max 120 points.
Fever | 4 weeks
  Incidence of infections with high fever (patients judgement)
CD16 | 4 weeks
  immunophenotyping of peripheral blood mononuclear cells (PBMCs) with measurement of soluble CD16
ADAM17 | 4 weeks
  immunophenotyping of peripheral blood mononuclear cells (PBMCs) with measurement of soluble ADAM17
transcriptomics | 4 weeks
  RNA sequencing for large-scale study of gene expression in circulation
microRNAs | 4 weeks
  large-scale study of microRNAs in circulation
proteomics | 4 weeks
  large-scale study of proteomes (proteins produced in study subjects)
metabolomics | 4 weeks
  large-scale study of metabolome (metabolites produced in study subjects)
hsCRP fibrinogen, immunoglobulin | 4 weeks
  High-sensitivity C-reactive Protein (laboratory measurement)
SR | 4 weeks
  erythrocyte sedimentation rate (laboratory measurement)
fibrinogen | 4 weeks
  fibrinogen (laboratory measurement)
immunoglobulins | 4 weeks
  immunoglobulin levels in fem klasser: IgA, IgD, IgE, IgG och IgM

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Chantzichristos, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No